CLINICAL TRIAL: NCT03588013
Title: Study of Environmental Enteropathy and Malnutrition in Pakistan
Acronym: SEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University of Virginia (Other); Children's Hospital Medical Center, Cincinnati (Other); Bill and Melinda Gates Foundation (Other); Washington University School of Medicine (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dr Syed Asad Ali, Associate Professor, Department of Pediatrics and Child Health, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3836-Ped-ERC-15
Record Dates: First submitted 2018-06-19; First posted 2018-07-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Malnutrition, Child; Enteropathy; Vaccine Response Impaired; Stunting; Gastrointestinal Disease
MeSH Terms: conditions — Child Nutrition Disorders; Intestinal Diseases; Growth Disorders; Gastrointestinal Diseases | interventions — Educational Status; Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Intervention Model Description: 1. Moderately or severely malnourished (weight for height Z score (WHZ) < -2) children
  2. Well-nourished (WHZ > 0) children
  3. Control group of children in the US with celiac disease
  4. Control group of children in the US with Crohn's disease
  5. Control group of healthy age-matched children in the US
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Moderate/severe malnourishment (Experimental): Pakistani children from age 0 to 6 months with weight for height Z score (WHZ) < -2 at the time of enrollment. Parents/caregivers of all participants will undergo a series of rehabilitative interventions to improve the child's nutrition and growth. Those participants who remain WHZ < -2 despite interventions are eligible for medical evaluation for more advanced workup of malnutrition, including UGI endoscopy and biopsy.
  Interventions: Other: Nutritional education; Dietary Supplement: Ready to Use Therapeutic Food; Procedure: Upper gastrointestinal endoscopy with biopsy
- Well nourished children (Active Comparator): Pakistani children from age 0 to 6 months who would be growing normally, with WHZ > 0, to serve as controls. Parents/caregivers of all participants will undergo a series of rehabilitative interventions to improve the child's nutrition and growth.
  Interventions: Other: Nutritional education
- US children with celiac disease (No Intervention): Comparative group for the Pakistani WHZ <-2 children who undergo UGI endoscopy and biopsy. Environmental Enteropathy and celiac disease have some shared features therefore we plan to enroll children under the age of 6 years with newly diagnosed celiac disease per endoscopy at CCHMC to assess the extent to which gene signatures and associated biologic pathways for children with celiac disease or environmental enteropathy overlap or differ.
- US children with Crohn's disease (No Intervention): Comparative group for the Pakistani WHZ <-2 children who undergo UGI endoscopy and biopsy. As some differentially expressed ileal gene signatures for Crohn's disease bear remarkable similarities to individual gene expression patterns previously reported for EE, children under the age of 10 years with newly diagnosed Crohn's disease per endoscopy at CCHMC will be enrolled to study these similarities and any differences
- Healthy age-matched US children (No Intervention): Comparative group for the Pakistani WHZ <-2 children who undergo UGI endoscopy and biopsy. Number of upper gastrointestinal endoscopies performed in children less than 2 years old are limited in Pakistan, therefore US age-matched controls will be used; healthy children < 3 years old will be enrolled, who will undergo endoscopy at CCHMC as part of a diagnostic workup for digestive symptoms, but whose biopsies and diagnoses are not supportive of eosinophilic esophagitis, celiac disease, or inflammatory bowel disease, and who were not treated with antibiotics ≤ 4 weeks prior to endoscopy.

INTERVENTIONS:
Other: Nutritional education — 4 week home delivered educational program that will focus on breast feeding and complimentary feeding. If child remains WHZ < -2 at by 9 months of age families will be shown 10 minute educational video detailing best practices for complimentary feeding.
  Other Names: Education
  Arms: Moderate/severe malnourishment; Well nourished children
Dietary Supplement: Ready to Use Therapeutic Food — If child remains WHZ < -2 despite nutritional education then will be managed according to Pakistan's Community Management of Acute Malnutrition protocol. This will include provision of ready to use therapeutic food (RUTF) to the child at home with close follow up. Utilization of the RUTF will be monitored closely by bi-weekly home visits.
  Other Names: RUTF
  Arms: Moderate/severe malnourishment
Procedure: Upper gastrointestinal endoscopy with biopsy — If child remains at WHZ < -2 despite educational and dietary interventions, then will undergo medical evaluation for assessment of need for more advanced workup of malnutrition, including UGI endoscopy at AKUH. Results of the advanced work up, including the UGI endoscopy, will guide future management of these children.
  Other Names: UGI endoscopy; Biopsy; Esophagoduodenoscopy
  Arms: Moderate/severe malnourishment

SUMMARY:
Environmental Enteropathy (EE) is an acquired sub-clinical inflammatory gut condition in which alterations in intestinal structure, function, and local and systemic immune activation lead to impaired vaccine responses, decreased cognitive potential and undernutrition in low-middle income countries. Approximately half of all global deaths in children aged less than five years are attributable to undernutrition making the study of EE an area of critical priority. However, given the operational limitations and ethical considerations for safely obtaining intestinal biopsies from young children in low resource settings, there have been few detailed investigations of human intestinal tissue in this vulnerable patient group for whom reversal of EE would provide the greatest benefit. EE biomarkers have been studied in different settings but these have not been correlated with the gold standard histopathology confirmation. The Study of Environment Enteropathy and Malnutrition in Pakistan (SEEM Pakistan) is designed to better understand the pathophysiology, predictors, biomarkers, and potential management strategies of EE to inform strategies to eradicate this debilitating pathology.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-6 months from Matiari, Pakistan with weight for height Z score (WHZ) < -2 at the time of enrollment
* Children aged 0 to 6 months from Matiari, Pakistan who would be growing normally, with WHZ > 0, to serve as controls
* Healthy control children under the age of 3 years, who will undergo endoscopy at CCHMC
* Children under the age of 6 years with newly diagnosed celiac disease per endoscopy at CCHMC
* Children under the age of 10 years with newly diagnosed Crohn's disease per endoscopy at CCHMC

Exclusion Criteria:

* For healthy control children < 3 years old undergoing endoscopy at CCHMC, biopsies and diagnoses should not supportive of eosinophilic esophagitis
* For healthy control children < 3 years old undergoing endoscopy at CCHMC, biopsies and diagnoses should not supportive of celiac disease
* For healthy control children < 3 years old undergoing endoscopy at CCHMC, biopsies and diagnoses should not supportive of inflammatory bowel disease
* For healthy control children < 3 years old undergoing endoscopy at CCHMC, children should not have been treated with antibiotics ≤ 4 weeks prior to endoscopy

Ages: 0 Days to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 416 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Nutritional status in children assessed by measuring parameters of growth at 3-6 months of age | Approximately 3-6 months after entry into study
  Our birth cohort will be assessed for nutritional status by measuring parameters of growth, length, weight and height. These measurements will be calculated as Z scores according to WHO tables and children will be divided into the appropriate categories: Stunting as Length for Age Z-score < -2 SD (standard deviation), underweight as Weight-for-Age Z-score < -2 SD and wasting as Weight-for-Length Z-score < -2 SD, or normal-for-age.
Nutritional status in children assessed by measuring parameters of growth at 9 months of age | At approximately 9 months after entry into study
  Our birth cohort will be assessed for nutritional status by measuring parameters of growth, length, weight and height. These measurements will be calculated as Z scores according to WHO tables and children will be divided into the appropriate categories: Stunting as Length for Age Z-score < -2 SD (standard deviation), underweight as Weight-for-Age Z-score < -2 SD and wasting as Weight-for-Length Z-score < -2 SD, or normal-for-age.
Association of biomarkers with Environmental Enteropathy at 3-6 months of age | Approximately 3-6 months after entry into study
  Serum, stool, and urine biomarkers of EE will be collected and tested in malnourished and well-nourished children
Association of biomarkers with Environmental Enteropathy at 9 months of age | At approximately 9 months after entry into study
  Serum, stool, and urine biomarkers of EE will be collected and tested in malnourished and well-nourished children
Association of biomarkers with Environmental Enteropathy at the time of endoscopy and biopsy | At approximately 15 months after entry into study
  Serum, stool, and urine biomarkers of EE will be collected and tested in those children who are eligible to undergo upper GI endoscopy and biopsy
The use of UGI biopsy tissue for histopathological and multiomic workup for validation of biomarkers associated with EE | At approximately 15 months after entry into study
  Biopsy specimens from UGI endoscopy obtained from eligible children will be used for detailed histopathologic and multiomic work up to study the pathophysiology of EE, validate current biomarkers, and generate novel biomarker candidates

CONTACTS AND LOCATIONS:
Overall Officials: Syed Asad Ali, MD, MPH, Principal Investigator — Aga Khan University; Sean R Moore, MD, Principal Investigator — University of Virginia
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed S, Iqbal J, Sadiq K, Umrani F, Rizvi A, Kabir F, Jamil Z, Syed S, Ehsan L, Zulqarnain F, Sajid M, Hotwani A, Rahman N, Ma JZ, McNeal M, Ann Costa Clemens S, Talat Iqbal N, Moore SR, Ali A. Association of Anti-Rotavirus IgA Seroconversion with Growth, Environmental Enteric Dysfunction and Enteropathogens in Rural Pakistani Infants. Vaccine. 2022 May 31;40(25):3444-3451. doi: 10.1016/j.vaccine.2022.04.032. Epub 2022 May 6. PMID 35534310
- [Derived] Zhao X, Setchell KDR, Huang R, Mallawaarachchi I, Ehsan L, Dobrzykowski Iii E, Zhao J, Syed S, Ma JZ, Iqbal NT, Iqbal J, Sadiq K, Ahmed S, Haberman Y, Denson LA, Ali SA, Moore SR. Bile Acid Profiling Reveals Distinct Signatures in Undernourished Children with Environmental Enteric Dysfunction. J Nutr. 2021 Dec 3;151(12):3689-3700. doi: 10.1093/jn/nxab321. PMID 34718665
- [Derived] Haberman Y, Iqbal NT, Ghandikota S, Mallawaarachchi I, Tzipi Braun, Dexheimer PJ, Rahman N, Hadar R, Sadiq K, Ahmad Z, Idress R, Iqbal J, Ahmed S, Hotwani A, Umrani F, Ehsan L, Medlock G, Syed S, Moskaluk C, Ma JZ, Jegga AG, Moore SR, Ali SA, Denson LA. Mucosal Genomics Implicate Lymphocyte Activation and Lipid Metabolism in Refractory Environmental Enteric Dysfunction. Gastroenterology. 2021 May;160(6):2055-2071.e0. doi: 10.1053/j.gastro.2021.01.221. Epub 2021 Jan 29. PMID 33524399
- [Derived] Iqbal NT, Syed S, Sadiq K, Khan MN, Iqbal J, Ma JZ, Umrani F, Ahmed S, Maier EA, Denson LA, Haberman Y, McNeal MM, Setchell KDR, Zhao X, Qureshi S, Shen L, Moskaluk CA, Liu TC, Yilmaz O, Brown DE, Barratt MJ, Kung VL, Gordon JI, Moore SR, Ali SA. Study of Environmental Enteropathy and Malnutrition (SEEM) in Pakistan: protocols for biopsy based biomarker discovery and validation. BMC Pediatr. 2019 Jul 22;19(1):247. doi: 10.1186/s12887-019-1564-x. PMID 31331393